CLINICAL TRIAL: NCT00276809
Title: Campath 1H (Alemtuzumab) Combined With High-Dose Therapy and Autologous Stem Cell Transplantation in Chronic Lymphocytic Leukemia
Brief Title: Combination Chemotherapy, Total-Body Irradiation, and Alemtuzumab in Treating Patients Undergoing an Autologous Stem Cell Transplant for Stage I, Stage II, Stage III, or Stage IV Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CLL3C; EU-20556; MEDAC-GCLLSG-CLL3C
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Filgrastim; Carmustine; Cyclophosphamide; Cytarabine; Dexamethasone; Etoposide; fludarabine phosphate; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: alemtuzumab
Biological: filgrastim
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide
Drug: fludarabine phosphate
Drug: melphalan
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving combination chemotherapy before a peripheral blood stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as G-CSF, and certain chemotherapy drugs, helps stem cells move from the bone marrow to the blood so they can be collected and stored. A monoclonal antibody, such as alemtuzumab, is given to kill any remaining cancer cells. Chemotherapy and radiation therapy (total-body irradiation) are given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy. Giving combination chemotherapy, total-body irradiation, and alemtuzumab together with autologous peripheral stem cell transplant may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with total-body irradiation and alemtuzumab works in treating patients undergoing an autologous stem cell transplant for stage I, stage II, stage III, or stage IV chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of cytoreductive fludarabine and cyclophosphamide followed by high-dose myeloablative therapy comprising total-body irradiation, cyclophosphamide, and alemtuzumab in patients undergoing autologous filgrastim (G-CSF)-mobilized peripheral blood stem cell transplantation for stage I-IV chronic lymphocytic leukemia.

Secondary

* Determine the clinical and molecular remission rate and duration in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter, open label, nonrandomized study. Patients are assigned to 1 of 2 cohorts according to time of enrollment.

* Cytoreductive induction therapy: All patients receive fludarabine IV and cyclophosphamide IV on days 1-3. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) or partial response (PR) proceed to stem cell mobilization. Patients with stage III or IV disease at this point are removed from study.
* Stem cell mobilization: All patients receive Dexa-BEAM comprising oral dexamethasone once daily on days 1-10; carmustine IV and melphalan IV on day 2; and cytarabine IV twice daily and etoposide IV once daily on days 4-7. Patients also receive filgrastim (G-CSF) subcutaneously beginning on day 8 and continuing until leukapheresis is completed. Patients undergo peripheral blood stem cell (PBSC) harvest between days 20 and 28. Patients without an adequate number of collected PBSCs may receive a second course of Dexa-BEAM. Patients achieving CR or very good PR proceed to high-dose myeloablative therapy and PBSC transplantation (PBSCT) with or without consolidation therapy.
* Consolidation therapy: Beginning between 1-2 months after completion of Dexa-BEAM, patients in cohort 2 receive alemtuzumab IV over 2 hours on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 and then proceed to high-dose myeloablative therapy and PBSCT within 1 month after completion of consolidation therapy. Patients in cohort 1 do not receive consolidation therapy and proceed directly to high-dose therapy within 3 months after completion of stem cell mobilization.
* High-dose myeloablative therapy and PBSCT: Patients undergo total-body irradiation on days -7 to -5. Patients then receive cyclophosphamide IV on days -4 and -3 and alemtuzumab IV over 2 hours on days -10, -9, -8, -6, and -4. Patients undergo PBSCT on day 0.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Chronic lymphocytic leukemia (CLL), meeting 1 of the following stage criteria:

  * Stage I-IV disease
  * Binet stage B or C disease
  * Binet stage A disease at high risk for rapid disease progression, as defined by both of the following criteria:

    * Nonnodular marrow infiltration and/or lymphocyte doubling time < 12 months
    * Thymidine kinase > 7.0 U/L and/or ß-2-microglobulin > 3.5 mg/L
* Polymerase chain reaction-amplifiable clonal CDR III rearrangement of the immunoglobulin variable heavy chain gene
* No Richter's syndrome or B-prolymphocytic leukemia

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* No concurrent disease resulting in major organ dysfunction
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other concurrent malignancy
* No New York Heart Association class III or IV cardiac failure
* No cardiomyopathy
* No history of myocardial infarction
* No symptomatic coronary heart disease
* No severe cardiac arrhythmia
* No severe or uncontrolled hypertension
* No chronic pulmonary disease
* No pulmonary function test impairment
* No severe or uncontrolled diabetes mellitus
* Bilirubin or transaminases ≤ 1.5 times upper limit of normal
* Creatinine ≤ 1.4 mg/dL
* No cerebral dysfunction
* No severe psychiatric impairment
* No drug addiction or alcoholism
* Negative HIV
* Negative Hepatitis B or C
* No allergy to any of the protocol drugs
* No history of anaphylactic reaction to monoclonal antibodies
* No active infection

PRIOR CONCURRENT THERAPY:

* No more than 1 prior chemotherapy regimen OR chemotherapy that lasted > 6 months
* No prior radiotherapy
* No prior treatment with alemtuzumab
* No prior long-term (> 1 month) systemic corticosteroids
* No prior therapy with dexamethasone, carmustine, etoposide, cytarabine, and melphalan (Dexa-BEAM)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-06; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of CAMPATH-1H included into the myeloablative regimen (cyclophosphamide and TBI) of the CLL3 protocol monitoring of treatment related mortality and morbidity (CTC scale) continuous

SECONDARY OUTCOMES:
Rate and duration of molecular responses MRD levels continuous
Rate and duration of clinical remissions NCIE sponsored remission criteria for CLL continuous
Overall survival time from treatment to death continuous

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Stilgenbauer, MD, Study Chair — Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm
Locations (12):
- Germany (12):
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Essen, Essen
  - Asklepios Klinik St. Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Universitatsklinik Mainz, Mainz
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm

REFERENCES:
- See also: German CLL Study Group — http://www.dcllsg.de